CLINICAL TRIAL: NCT04078763
Title: Rehabilitation of the Auditory Space for Bilateral Cochlear Implant Users : a Feasibility Study
Acronym: RECOVER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69HCL19_0238
Record Dates: First submitted 2019-09-02; First posted 2019-09-06 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Cochlear Prosthesis Implantation
Keywords: Spatial hearing perception; cochlear prosthesis implantation users; virtual reality; rehabilitation
MeSH Terms: interventions — Feedback, Sensory; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- visual-auditory feedback (Experimental): Patients included in this arm will follow the rehabilitation protocol with visual-auditory feedback. Performance of the rehabilitation protocol will be assessed thanks to 3 tests : SPHERE protocol, French Matrix Test and SSQ15 questionnaire
  Interventions: Behavioral: Rehabilitation protocol with visual-auditory feedback; Behavioral: SPHERE protocol; Behavioral: French Matrix Test; Behavioral: Speech Spatial and Qualities of Hearing Scale (SSQ15) questionnaire
- visual feedback (Experimental): Patients included in this arm will follow the rehabilitation protocol with visual feedback. Performance of the rehabilitation protocol will be assessed thanks to 3 tests : SPHERE protocol, French Matrix Test and SSQ15 questionnaire
  Interventions: Behavioral: Rehabilitation protocol with visual feedback; Behavioral: SPHERE protocol; Behavioral: French Matrix Test; Behavioral: Speech Spatial and Qualities of Hearing Scale (SSQ15) questionnaire

INTERVENTIONS:
Behavioral: Rehabilitation protocol with visual-auditory feedback — The rehabilitation protocol with visual-auditory feedback is based on 8 sessions, over a period of 1 month, with 2 sessions per week. Each session lasts 45 minutes. During a session, the participant has to localize a sound around him, at hand. For this, he has to direct his head (which acts as a pointer) to the place where he seems to get the sound. Then, he validates his answer using the joystick placed in his hand. Regardless of the answer given (exact or incorrect), the subject will always have a visual-auditory feedback
  Arms: visual-auditory feedback
Behavioral: Rehabilitation protocol with visual feedback — The rehabilitation protocol with visual feedback is based on 8 sessions, over a period of 1 month, with 2 sessions per week. Each session lasts 45 minutes. During a session, the participant has to localize a sound around him, at hand. For this, he has to direct his head (which acts as a pointer) to the place where he seems to get the sound. Then, he validates his answer using the joystick placed in his hand. Regardless of the answer given (exact or incorrect), the subject will only have a visual feedback.
  Arms: visual feedback
Behavioral: SPHERE protocol — Data from spatial sound perception will be recorded in three dimensional space (azimuth, elevation, and depth). First, the pointing error will be computed separately for azimuth, elevation, and depth, in terms of constant error (absolute and signed) and variable error. Then, these separate errors will be combined into a cumulative error "3d-D", hence summarizing all three space dimensions, and taking into account absolute and variable error in one measure. This lasts 10 minutes and the result is expressed by the 3d-D value
Behavioral: French Matrix Test — This test assesses the intelligibility threshold defined as the noise level (in decibels) for which the subject can repeat 50% of the words heard (in dichotic listening), resulting in an Speech Recognition Threshold (SRT) value. This test lasts 10 minutes.
Behavioral: Speech Spatial and Qualities of Hearing Scale (SSQ15) questionnaire — 15 items questionnaire (each answer to questions is quoted between 0 and 10) resulting in a global SSQ 15 score. It takes 10 minutes to fill the questionnaire.

SUMMARY:
A new Neuro-Immersion system based on virtual reality and 3D motion tracking has been developed recently, allowing to evaluate and record the spatial localization performance of cochlear implant (CI) users. This system allows to highlight localization deficits in three-dimensional space for all CI patients. Unfortunately, there is currently no suitable postoperative management for these localization problems. However, the discomfort felt by patients is clearly verbalized. Thanks to the new virtual reality system, it is now possible to develop a rehabilitation protocol adapted to each patient. This project will focus on the evaluation of a spatial auditory rehabilitation, based on unisensory (visual) or multisensory (auditory and visual) feedback, for bilateral CI adults.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years inclusive
* Use of the second CI for at least 1 year
* Regular follow-up in the Ear Nose and Throat department of Edouard Herriot Hospital in Lyon
* Post-lingual deafness
* Average voice recognition over 80% with 2 Cochlear Implants
* Normal vision (with or without correction)
* Able to understand the experimental instructions
* Affiliated to a social security scheme

Exclusion Criteria:

* Oculomotor disorder
* Bilateral vestibular areflexia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2020-09-04 (Actual); Study Completion 2020-09-04 (Actual)

PRIMARY OUTCOMES:
Short term rehabilitation effect on the spatial auditory performance - 4 sessions | 4 weeks after inclusion
  This effect will be defined as any change in auditory performance scores (3d-D value OR SRT value or SSQ15 questionnaire score) between baseline (before rehabilitation starts) and short term rehabilitation (4 rehabilitation sessions)
Short term rehabilitation effect on the spatial auditory performance - 8 sessions | 6 weeks after inclusion
  This effect will be defined as any change in auditory performance scores (3d-D value OR SRT value or SSQ15 questionnaire score) between baseline (before rehabilitation starts) and short term rehabilitation (8 rehabilitation sessions)

SECONDARY OUTCOMES:
Percentage of sessions performed on all the rehabilitation sessions during the protocol | 6 weeks after inclusion
  compliance of participant to attend the rehabilitation sessions will be measured by calculating the percentage of sessions performed on all the rehabilitation sessions during the protocol
Middle term rehabilitation effect on the spatial auditory performance | 10 to 12 weeks after inclusion
  This effect will be defined as any change in auditory performance scores (3d-D value or SRT value or SSQ15 questionnaire score) between baseline (before rehabilitation starts) and 8 to 10 weeks after the first rehabilitation session
Measure of auditory performance tests own effect | 2 weeks after inclusion
  This effect corresponds to the difference between auditory performance scores (3d-D value, SRT value and SSQ15 questionnaire score) at inclusion and 2 weeks after inclusion, before rehabilitation starts.
Short term feedback effect on spatial auditory performance | 4 weeks after inclusion
  The short term feedback effect on spatial auditory performance will be assessed by comparing the auditory performance scores (3d-D value, SRT value and SSQ15 questionnaire score) of the two groups after 4 rehabilitation sessions
Short term feedback effect on spatial auditory performance | 6 weeks after inclusion
  The short term feedback effect on spatial auditory performance will be assessed by comparing the auditory performance scores (3d-D value, SRT value and SSQ15 questionnaire score) of the two groups after 8 rehabilitation sessions
Middle term feedback effect on spatial auditory performance | 10 to 12 weeks after inclusion
  The middle term feedback effect on spatial auditory performance will be assessed by comparing the auditory performance scores (3d-D value, SRT value and SSQ15 questionnaire score) of the two groups 8 to 10 weeks after the first rehabilitation session

CONTACTS AND LOCATIONS:
Overall Officials: Eric TRUY, Professor, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Edouard Herriot, Lyon, France

REFERENCES:
- [Result] Coudert A, Verdelet G, Reilly KT, Truy E, Gaveau V. Intensive Training of Spatial Hearing Promotes Auditory Abilities of Bilateral Cochlear Implant Adults: A Pilot Study. Ear Hear. 2023 Jan-Feb 01;44(1):61-76. doi: 10.1097/AUD.0000000000001256. Epub 2022 Aug 9. PMID 35943235